CLINICAL TRIAL: NCT00243464
Title: Calcipotriol Plus Betamethasone Dipropionate Gel Compared to DAIVONEX/DOVONEX Scalp Solution in Patients With Scalp Psoriasis
Brief Title: Efficacy of Calcipotriol Plus Betamethasone Gel Versus Calcipotriol Scalp Solution in Scalp Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBL 0503 INT
Record Dates: First submitted 2005-10-21; First posted 2005-10-24 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2015-03

CONDITIONS: Psoriasis of Scalp
MeSH Terms: interventions — calcipotriene; betamethasone-17,21-dipropionate

INTERVENTIONS:
Drug: Calcipotriol plus betamethasone dipropionate (LEO80185 gel)

SUMMARY:
The purpose of this study is to evaluate whether once daily treatment for up to 8 weeks of calcipotriol plus betamethasone dipropionate gel is more effective than twice daily treatment of calcipotriol scalp solution in patients with scalp psoriasis. The primary outcome is patients with clear or minimal disease after 8 weeks treatment.

Further the occurrence of relapse and rebound after end of treatment in patients with clear or minimal disease will be investigated.

ELIGIBILITY:
Main Inclusion Criteria:

* Scalp psoriasis amenable to topical treatment
* Psoriasis vulgaris on trunk and/or limbs
* Extent of scalp psoriasis involving more than 10% of the total scalp area
* Disease severity on the scalp graded as moderate or worse by the investigator
* Consenting out-patients of 18 years or above

Main Exclusion Criteria:

* PUVA or Grenz ray therapy within 4 weeks prior to randomisation
* UVB therapy within 2 weeks prior to randomisation
* Systemic treatment with biological therapies, with a possible effect on scalp psoriasis within 6 months prior to randomisation
* Systemic treatment with all other therapies than biologicals, with a possible effect on scalp psoriasis (e.g., corticosteroids, vitamin D analogues, retinoids, immunosuppressants) within 4 weeks prior to randomisation
* Any topical treatment of the scalp (except for non steroid medicated shampoos and emollients) within 2 weeks prior to randomisation
* Topical treatment of the face, trunk and/or limbs with very potent WHO group IV corticosteroids within 2 weeks prior to randomisation
* Current diagnosis of erythrodermic, exfoliative or pustular psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-09; Study Completion 2006-05

PRIMARY OUTCOMES:
Overall disease severity according to investigator's assessment at week 8

SECONDARY OUTCOMES:
Total sign score at week 8
Score for redness, thickness and scaliness at week 8
Overall disease severity according to the investigator's assessment at week 2 and 4
Overall disease severity according to patients at week 8
Relapse and rebound during the study

CONTACTS AND LOCATIONS:
Overall Officials: Knud Kragballe, MD, Principal Investigator — Department of Dermatology, Marselisborg Centres
Locations (5):
- Universitair Ziekenhuis Sint Raphaël, Dienst Dermatologie, Leuven, Belgium
- Windsor Clinical Research Inc., Windsor, Ontario, Canada
- Department of Dermatology, Marselisborg Centres, Aarhus, Denmark
- Hôpital de L'Archet, Service de Dermatologie, Nice, France
- Läkarhuset, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en